CLINICAL TRIAL: NCT04447716
Title: A Phase I Study of Venetoclax + Lenalidomide + Rituximab Hyaluronidase in Relapsed or Refractory (R/R) Indolent Non-Hodgkin's Lymphoma (iNHL).
Brief Title: An Early Phase Study of Venetoclax, Lenalidomide, and Rituximab/Hyaluronidase in Slow-Growing Lymphomas That Have Come Back After Treatment or Have Not Responded to Treatment
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19P.835; JT 14408 (Other: JeffTrial Number)
Record Dates: First submitted 2020-04-09; First posted 2020-06-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Follicular Lymphoma; Recurrent Indolent Adult Non-Hodgkin Lymphoma; Recurrent Marginal Zone Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Follicular Lymphoma; Refractory Indolent Adult Non-Hodgkin Lymphoma; Refractory Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — venetoclax; Lenalidomide; Rituximab; CT-P10; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (venetoclax, lenalidomide, rituximab, hyaluronidase) (Experimental): Patient receive venetoclax PO QD on days 1-28. Beginning cycle 2, patients receive lenalidomide PO QD on days 1-21. Patients also receive rituximab IV on days 1, 8, 15, and 22 of cycle 2 and rituximab hyaluronidase (if no significant infusion reaction to rituximab) SC on day 1 of cycles 4, 6, 8, 10, and 12. Patients may receive rituximab IV (instead of rituximab hyaluronidase) on days 1, 8, 15, and 22 of cycles 4, 6, 8, 10, and 12 if the patient requires rituximab IV in the opinion of the treating physician. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Venetoclax; Drug: Lenalidomide; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human

INTERVENTIONS:
Drug: Venetoclax — Given PO
  Other Names: 1257044-40-8,; 4-(4-((2-(4-Chlorophenyl)-4; 4-dimethylcyclohex-1-en-1-yl)methyl)piperazin-1-yl)-N-((3-nitro-4-((tetrahydro-2H-pyran-4-ylmethyl)amino)phenyl)sulfonyl)-2-(1H-pyrrolo(2,3-b)pyridin-5-yloxy)benzamide,; ABT-0199,; ABT-199,; ABT199,; RG7601,; GDC-0199,
Drug: Lenalidomide — Given PO
  Other Names: 191732-72-6,; 3-(4-Amino-1-oxo-1,3-dihydro-2H-isoindol-2-yl)piperidine-2,6-dione,; 703813,; CC-5013; Revlimid; CC5013; CDC 501,; lenalidomide,
Biological: Rituximab — Given IV
  Other Names: 174722-31-7,; 687451,; ABP 798,; BI 695500,; C2B8 Monoclonal Antibody,; Chimeric Anti-CD20 Antibody,; CT-P10,; IDEC-102,; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody,; MabThera,; Monoclonal Antibody IDEC-C2B8,; PF-05280586,; Rituxan,; Rituximab,; RITUX
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela,; Rituximab Plus Hyaluronidase,; Rituximab/Hyaluronidase,; Rituximab/Hyaluronidase Human

SUMMARY:
This phase I trial studies the side effects and best dose of venetoclax when given together with lenalidomide and rituximab hyaluronidase in treating patients with follicular lymphoma and marginal zone lymphoma that has come back after treatment (relapsed) or has not responded to treatment (refractory). Venetoclax may stop the growth of cancer cells by blocking the action of a protein called Bcl-2, that helps cancer cells survive. Immunotherapy with lenalidomide, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Immunotherapy with monoclonal antibodies, such as rituximab and rituximab hyaluronidase, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The purpose of this research is to determine if the combination of three drugs, venetoclax, lenalidomide, and rituximab hyaluronidase are safe to administer in patients whose low-grade lymphoma (follicular or marginal zone) has come back after initial therapy or was not responsive to initial therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety (and the recommended phase 2 dose [RP2D]), of the combination of venetoclax, lenalidomide, and rituximab hyaluronidase in patients with relapsed/refractory (R/R) follicular lymphoma (FL) and marginal zone lymphoma (MZL).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) with rituximab hyaluronidase, venetoclax, and lenalidomide.

II. To determine the 2-year progression-free survival (PFS) with rituximab hyaluronidase, venetoclax, and lenalidomide.

III. To determine the overall survival (OS) following therapy with rituximab hyaluronidase, venetoclax, and lenalidomide.

CORRELATIVE STUDY OBJECTIVES:

I. Describe changes in the level of expression and expression ratio between anti-apoptotic and pro-apoptotic BCL-2 family members before and after therapy with venetoclax/lenalidomide/rituximab hyaluronidase for each patient.

II. Examine the metabolic landscape before and after venetoclax/lenalidomide/rituximab hyaluronidase and their effects on mitochondrial metabolism.

III. Describe the immune effects of venetoclax and its effects on serum cytokines and different immune cell subsets (e.g. B-cells, T-cells, dendritic cells, etc.) in addition to T-cell activation markers and expression of immune checkpoint proteins.

OUTLINE: This is a dose-escalation study of venetoclax.

Patient receive venetoclax orally (PO) once daily (QD) on days 1-28. Beginning cycle 2, patients receive lenalidomide PO QD on days 1-21. Patients also receive rituximab intravenously (IV) on days 1, 8, 15, and 22 of cycle 2 and rituximab hyaluronidase (if no significant infusion reaction to rituximab) subcutaneously (SC) on day 1 of cycles 4, 6, 8, 10, and 12. Patients may receive rituximab IV (instead of rituximab hyaluronidase) on days 1, 8, 15, and 22 of cycles 4, 6, 8, 10, and 12 if the patient requires rituximab IV in the opinion of the treating physician. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent form

* Ability and willingness to comply with the requirements of the study protocol
* Able to swallow oral medications whole
* Patients must have received at least one prior systemic therapy
* Histologically confirmed indolent B-cell non-Hodgkin's lymphoma (NHL) of any of the following subtypes recognized by the World Health Organization (WHO) classification: Follicular lymphoma and marginal zone lymphoma. Patients with indolent non-Hodgkin's Lymphoma (iNHL) should have received at least 1 previous prior therapy
* Patients must have an indication for treatment by Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria in the opinion of the investigator
* Radiographically measurable disease by computed tomography (CT) scan, defined as at least one node > 1.5 cm in size
* All study participants must be registered into the mandatory lenalidomide risk evaluation and mitigation strategy (REMS) program, and be willing and able to comply with the requirements of the REMS program
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the lenalidomide REMS program
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. Patients intolerant to aspirin (ASA) may use low molecular weight heparin or equivalent. Inability to take any form of prophylaxis excludes participation
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Hemoglobin >= 9 g/dL (unless caused by underlying disease, as established by extensive bone marrow involvement or as a result of hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator)
* Absolute neutrophil count >= 1.0 x 10^9/L (unless caused by underlying disease, as established by extensive bone marrow involvement or as a result of hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator)
* Platelet count >= 75 x 10^9/L (unless caused by underlying disease, as established by extensive bone marrow involvement or as a result of hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator)
* International normalized ratio > 1.5 x upper limit of normal (ULN) for patients not receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) or activated PTT (aPTT) =< 1.5 x ULN
* Creatinine clearance >= 60 mL/min, calculated with the use of the 24-hour creatinine clearance or modified Cockcroft-Gault equation
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x ULN
* Total bilirubin =< 1.5 x ULN (or =< 3 x ULN for patients with documented Gilbert syndrome)
* Women of childbearing potential must have a negative serum or urine pregnancy test result within 14 days prior to registration
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 30 days after the last dose of venetoclax and lenalidomide or 12 months after the last dose of rituximab, whichever is longer * Women must refrain from donating eggs during this same period

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus) * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of rituximab and for at least 30 days after the last dose of venetoclax and lenalidomide whichever is longer. Men must refrain from donating sperm during this same period * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of rituximab to avoid exposing the embryo * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

Known hypersensitivity to any of the study drugs study drugs

* Known central nervous system (CNS) involvement by lymphoma
* Prior allogeneic stem cell transplant is not permitted if patient is fewer than 4 months from transplant and has either active graft versus host disease or on immunosuppression
* History of severe allergic reactions to humanized monoclonal antibodies
* Prior use of lenalidomide or venetoclax or other BCL2 family inhibitors; prior rituximab is allowed as long as they continue to express CD20 and are not rituximab refractory as defined as: * Did not respond (at least a partial response [PR]) to rituximab or rituximab (R)-chemoregimen therapy * Time to disease progression < 6 months after last rituximab dose
* History of other malignancy that could affect compliance with the protocol or interpretation of results * Patients with a history of curatively treated basal or squamous cell carcinoma or stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible * Patients with a malignancy that has been treated with surgery alone with curative intent will also be excluded. Individuals in documented remission without treatment for >= 2 years prior to enrollment may be included at the discretion of the investigator
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient, including renal disease that would preclude chemotherapy administration or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to registration
* Requires the use of warfarin (because of potential drug-drug interactions that may potentially increase the exposure of warfarin)
* Received the following agents within 7 days prior to registration: * Steroid therapy for anti-neoplastic intent * Strong and moderate CYP3A inhibitors * Strong and moderate CYP3A inducers * Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of venetoclax
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody * Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation * Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV deoxyribonucleic acid (DNA) is undetectable. These patients must be willing to undergo monthly DNA testing.
* Known infection with human immunodeficiency virus (HIV) or human T-cell leukemia virus 1 (HTLV-1)
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
* Pregnant or lactating, or intending to become pregnant during the study
* Recent major surgery (within 6 weeks prior to the start of cycle 1, day 1) other than for diagnosis
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Known allergy to both xanthine oxidase inhibitors and rasburicase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities | During the first 56 days of therapy
  Toxicity incidences assessed and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0, will be tabulated by patient cohort.

SECONDARY OUTCOMES:
Overall response rate | At the end of 12 month treatment period
  Defined as the sum of the proportions of patients achieving a complete (CR) or partial response (PR) according to the Lugano Response Criteria. Analyses of efficacy outcomes will be descriptive. A 90% confidence interval will be computed for the best response rate (CR+PR rate) during the 12 month treatment period.
Progression-free survival (PFS) | Time from study registration to documented disease progression or death from any cause, assessed at 2 years
  PFS distributions will be estimated using the Kaplan-Meier method, and the median PFS along with its corresponding 95% confidence interval will be reported.
Overall survival (OS) | Time from study registration to death from any cause, assessed at 2 years
  OS distributions will be estimated using the Kaplan-Meier method, and the median OS along with its corresponding 95% confidence interval will be reported.

OTHER OUTCOMES:
Level of expression and expression ratio between anti-apoptotic and pro-apoptotic BCL-2 family proteins measured by flow cytometry and messenger ribonucleic acid (mRNA) | 42 days of starting treatment through end of treatment
Metabolic landscape | 42 days of screening through until end of treatment
  Adenosine triphosphate (ATP) will be measured by mass spectroscopy and metabolic proteins will described by immunohistochemistry.
Immune profile | 42 days of starting treatment through until end of treatment
  Flow cytometry will be used to measure T-cell and B-cell subsetswill be used to quantitate PD-1/PD-L1.
Immune profile | 42 days of starting treatment through until end of treatment
  Immunohistochemistry will be used to quantitate PD-1/PD-L1.

CONTACTS AND LOCATIONS:
Overall Officials: Ubaldo R Martinez-Outschoorn, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States